CLINICAL TRIAL: NCT00697463
Title: Teriparatide for the Treatment of Idiopathic Osteoporosis in Premenopausal Women
Brief Title: Forteo for the Treatment of Unexplained Osteoporosis in Premenopausal Women
Acronym: IOPForteo
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Elizabeth Shane, Professor of Medicine, Endocrinology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAC6871
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Menopause; Fracture; Osteoporosis
Keywords: Teriparatide; Forteo; Osteopenia; Osteoporosis; Fracture; Low Bone Density; Premenopausal women
MeSH Terms: conditions — Fractures, Bone; Osteoporosis; Bone Diseases, Metabolic | interventions — Teriparatide; Parathyroid Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Women with Idiopathic osteoporosis (IOP) (Experimental): Each subject will receive 20 micrograms of Teriparatide (PTH 1-34) subcutaneously daily for 18 -24 months
  Interventions: Drug: Teriparatide (PTH 1-34)

INTERVENTIONS:
Drug: Teriparatide (PTH 1-34) — 20 micrograms subcutaneous injection daily
  Other Names: Forteo

SUMMARY:
Idiopathic osteoporosis (IOP) is an uncommon disorder in which otherwise healthy young individuals sustain one or more low-trauma fractures. Teriparatide [PTH(1-34)], which is FDA approved for treatment of osteoporosis in men and postmenopausal women, works by stimulating bone formation. The investigators hypothesize that teriparatide will significantly increase bone density (BMD) and improve bone structure in premenopausal women with IOP.

DETAILED DESCRIPTION:
Idiopathic osteoporosis (IOP) is an uncommon disorder in which otherwise healthy young individuals sustain one or more low-trauma fractures. In studies of IOP in men, histomorphometric indices of bone formation are depressed, and affected men respond to PTH(1-34) with robust increases in lumbar spine (LS) bone mineral density (BMD). This is the beginning of the third year of an R01 (AR4989603) investigating the etiology and pathogenesis, as well as the histomorphometric and bone microarchitectural features of IOP in premenopausal women. There is evidence of markedly decreased bone formation and microarchitectural deterioration with decreased mechanical competence/strength.

Teriparatide [PTH(1-34)] is an anabolic agent that stimulates bone formation and improves bone microarchitecture. Based on findings, the investigators hypothesize that teriparatide will significantly increase BMD and improve microarchitecture in premenopausal women with IOP.

This is an open-label study of carefully characterized premenopausal women with IOP who are participating in a NIH-funded study and who have fragility fractures or very low bone density. Participants in the study will receive 18-24 months of teriparatide and the effects on BMD and microstructure, bone mechanical competence, and bone turnover will be assessed. In order to assess whether teriparatide stimulates bone formation to the same extent in women with IOP as it does in normal women, the study will compare the short-term changes (2 and 4 weeks) in biochemical markers of bone formation in response to teriparatide between women with IOP and normal women who are participating in another NIH-funded study as controls.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women of all races.
* Ages 20 to 48.
* Regular menses (at least 8 periods in the last 12 months).
* FSH < 20 mIU/ml during the early follicular phase, to exclude women in the perimenopause.
* Fracture subjects: documented low trauma fracture(s) at age >= 18 (e.g., fracture associated with a fall from a standing height or less).
* Low BMD subjects: DXA BMD T score less than or equal to 2.5 at the LS, total hip, femoral neck or distal radius, who have not had a fracture.
* Control subjects: DXA BMD T score greater than or equal to 1.0 at the LS, total hip, femoral neck and distal radius, who have not had a fracture.
* All subjects must use appropriate birth control methods to prevent pregnancy for the duration of teriparatide treatment.

Exclusion Criteria:

* Secondary Causes of Osteoporosis.
* Disorders of mineral metabolism: primary or secondary hyperparathyroidism (serum intact PTH > 65 pg/ml), vitamin D deficiency (serum 25OHD < 30 ng/ml), hypercalciuria (>300 mg/g creatinine), Paget's disease, clinical osteomalacia, osteogenesis imperfecta (OI).
* Recent pregnancy or lactation (within past year).
* Prolonged amenorrhea (> 6 months) during reproductive years (except during pregnancy or lactation).
* History of anorexia nervosa.
* Malignancy, except cured basal or squamous cell skin carcinoma.
* Endocrinopathy: hyperthyroidism (elevated serum thyroxine and/or suppressed TSH), untreated hypothyroidism, Cushing's syndrome, prolactin-secreting pituitary adenoma.
* Renal insufficiency (serum creatinine above upper limit of female normal range).
* Liver disease (AST, ALT, bilirubin, total alkaline phosphatase activity above upper normal limit).
* Intestinal disorders (celiac disease, pancreatic insufficiency, inflammatory bowel disease).
* History or current use of glucocorticoids, anticonvulsants, anticoagulants, diuretics, methotrexate.
* Current use of depot preparations of progesterone or GnRH agonists.
* Current use of drug therapies for osteoporosis (estrogen preparations other than contraceptives, raloxifene, bisphosphonates, calcitonin, PTH). Subjects who agree to discontinue use of these medications will be eligible to participate 6 months after discontinuing raloxifene or calcitonin, and 12 months after discontinuing bisphosphonates. Total exposure to bisphosphonates must be < 1 year. Subjects who have taken PTH at any time in the past will not be eligible.
* Additional contraindications to teriparatide use: Unexplained elevated total or bone specific alkaline phosphatase or prior external beam or implant radiation therapy involving the skeleton.

Ages: 20 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08-20 (Actual); Primary Completion 2012-01-03 (Actual); Study Completion 2012-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shane, MD, Principal Investigator — Columbia University; Adi Cohen, MD, Study Director — Columbia University
Locations (2):
- United States (2):
  - Creighton University, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Premenopausal women, aged 20-48, with documented adult low trauma fractures or low aBMD by DXA; T score<-2.5 or Z score<-2.0 at the spine or hip and no history of adult low trauma fracture, were recruited at Columbia University Medical Center, NY and Creighton University, NE by advertisement, self- or physician referral.
Pre-assignment Details: No pre-assignment details to report
Groups:
- Women With Idiopathic Osteoporosis (IOP): Each subject will receive 20 micrograms of teriparatide subcutaneously daily.
  Teriparatide (PTH 1-34): 20 micrograms subcutaneous injection daily for 18- 24 months
Period: Overall Study
Arm/Group | Women With Idiopathic Osteoporosis (IOP)
Started | 22
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Women With Idiopathic Osteoporosis (IOP): Each subject will receive 20 micrograms of teriparatide subcutaneously daily.
  Teriparatide (PTH 1-34): 20 micrograms subcutaneous injection daily for 18-24 months
Arm/Group | Women With Idiopathic Osteoporosis (IOP)
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Lumbar Spine Bone Density by Dual Energy X-ray Absorptiometry (DXA)
Description: Areal BMD at the lumbar spine was measured by dual energy x-ray absorptiometry (DXA) at baseline and at 6, 12, 18, and 24 months, if possible.
Time Frame: Baseline, Month 18 or 24 reported
Population: Of 22 women with IOP who enrolled, one withdrew for personal reasons, therefore the overall number of participants analyzed is 21. The percentage of BMD change is calculated for each participant between baseline and Month 24 or between baseline and Month 18, whichever is the longer reported timeframe as some are lost to follow up by Month 24.
Measure: Mean (Standard Deviation); unit: percentage of BMD change
Arm/Group | Women With Idiopathic Osteoporosis (IOP)
Number analyzed (Participants) | 21
percentage of BMD change | 10.8 (8.3)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed through study completion.
Description: The definition of adverse event and/or serious adverse event used to collect adverse event information is the same.
Arm/Group | Women With Idiopathic Osteoporosis (IOP)
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 8/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women With Idiopathic Osteoporosis (IOP) (N=21)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1) — One participant had a single episode of hypercalcemia (serum calcium > 10.2 mg/dL) that resolved after per protocol reduction of calcium supplements.
Hypercalciuria (Renal and urinary disorders) | 6 (7) — 6 participants had 7 episodes of hypercalciuria (.300 mg/g creatinine) that resolved after per protocol reduction of calcium supplements.
Distal radius fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — One participant sustained a distal radius fracture after falling from a stool during the second 12 months.

LIMITATIONS AND CAVEATS:
Without an untreated control group, we cannot attribute the observed effects to teriparatide with certainty. The effects of teriparatide on fractures could not be evaluated. Six women received teriparatide for 18 months rather than for 24 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No